CLINICAL TRIAL: NCT06966986
Title: Radiofrequency-responsive Layered Double Hydroxides for Enhanced Arterial Embolization and Thermal Immunotherapy in Hepatocellular Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2024-140
Record Dates: First submitted 2024-11-25; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Liver Carcinoma
Keywords: Indocyanine green (ICG), radiofrequency ablation, microwave ablation, laparoscopy, liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- treatment after RFA: These samples will be used to assess the state of the patient's immune response, focusing on the following areas: Immune cell subpopulation analysis: Analysis is performed by flow cytometry to detect changes in the proportion of different immune cell subpopulations, specifically the number and functional status of CD8+ T cells, regulatory T cells (Tregs), and NK cells. Simulated radiofrequency ablation was performed in vitro, focusing on changes in the ablation range.

SUMMARY:
Liver cancer is one of the most common malignant tumors and the third leading cause of cancer-related deaths globally. Recent epidemiological studies show that in China, liver cancer ranks fourth in incidence and second in mortality among malignant tumors, posing a serious threat to human health. The common risk factors for liver cancer are chronic inflammatory infections caused by hepatitis B virus (HBV) and hepatitis C virus (HCV), which lead to liver cirrhosis and eventually develop into liver cancer.

The field of liver cancer treatment is characterized by its multidisciplinary approach and the coexistence of various therapeutic methods. Common treatment modalities include liver resection, liver transplantation, ablation therapies, and transcatheter arterial chemoembolization (TACE). Selecting appropriate treatment strategies based on the different stages of liver cancer can maximize therapeutic outcomes.

Although surgical intervention is considered the first-line curative treatment for liver cancer, a significant number of patients are unable to tolerate surgery due to varying degrees of liver cirrhosis and impaired liver function. The limited availability of treatment options results in a relatively low 5-year survival rate of approximately 18% for liver cancer patients. Liver cancer is insidious in onset, highly malignant, and progresses rapidly. Most patients are diagnosed at an advanced stage, having missed the optimal window for surgical resection.

For these patients, interventional therapies based on transcatheter arterial embolization (TAE) have shown excellent antitumor effects and are gradually becoming essential treatment methods for advanced liver cancer. In TAE, embolic agents are injected into the tumor's supplying arteries via a catheter to block the tumor's oxygen and nutrient supply. Currently, embolic agents primarily include liquid embolics (e.g., lipiodol) and solid agents (e.g., microspheres).

However, as a palliative treatment, TAE struggles to completely suppress tumor growth. This limitation arises because these embolic agents are unable to fully and permanently block all tumor vasculature, allowing tumors to establish collateral circulation after the procedure. Additionally, the hypoxic tumor microenvironment created post-procedure stimulates rapid proliferation of liver cancer cells. Consequently, it is critical to develop effective strategies to improve the outcomes of TAE.

Radiofrequency ablation (RFA), a common thermal ablation method for liver cancer in clinical practice, has been widely applied. Leading medical associations, including the U.S. National Comprehensive Cancer Network (NCCN) and the Asia-Pacific Association for the Study of the Liver (APASL), have recognized RFA as a first-line treatment for solitary liver tumors ≤3 cm in size.

During RFA, the central region of the tumor reaches temperatures above 50°C, inducing coagulative necrosis of solid tumors, while the surrounding area, referred to as the transition zone, experiences sublethal heat stress. However, incomplete radiofrequency ablation (iRFA) can occur due to factors such as large tumor size, thermal sink effects of blood vessels, and undetected micro-satellite lesions, leading to rapid recurrence or metastasis of residual tumor tissue.

Studies have reported that RFA can induce specific immune responses by releasing tumor-associated antigens, damage-associated molecular patterns (DAMPs), and pro-inflammatory cytokines from denatured tumor cells. However, the antitumor immune response elicited by RFA is often transient and weak. Moreover, it may trigger a series of immunosuppressive responses, further complicating the overall therapeutic outcome.

ELIGIBILITY:
Inclusion Criteria:

* individual tumors were less than 5 cm in diameter. The number of multiple tumors was not more than 3, and the diameter of each tumor was not more than 3 cm, and there was no extrahepatic metastasis. Child-Pugh A or B; There is no refractory ascites or irremediable coagulation dysfunction; Prothrombin activity higher than 40%, platelet count more than 500,000/L; RFA with healing purpose.

Exclusion Criteria:

* presence of vascular infiltration and extrahepatic metastasis; Severe clotting disorders; Severe cardiopulmonary insufficiency or uncontrolled liver decompensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical data of patients undergoing radiofrequency ablation of liver cancer in the Fourth Affiliated Hospital of Zhejiang University were collected
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Immune | 2024-2026
  Changes in the proportion of different immune cell subsets were detected, especially the number and functional status of CD8+ T cells, regulatory T cells (Tregs), and NK cells

SECONDARY OUTCOMES:
Immune | 2024-2026
  IFN-γ

OTHER OUTCOMES:
Immune | 2024-2026
  RNA-sequency

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No